CLINICAL TRIAL: NCT00353197
Title: The Derivation of New Human Embryonic Stem Cell Lines for Clinical Use
Brief Title: Derivation of New Human Embryonic Stem Cell Lines Lines for Clinical Use
Status: Recruiting | Type: Observational
Sponsor: Hadassah Medical Organization (Other)
Responsible Party: Sponsor
Other Study IDs: 33-26.07.02-HMO-CTIL
Record Dates: First submitted 2006-07-16; First posted 2006-07-18 (Estimated); Last update posted 2025-03-05 (Actual); Status verified 2025-03

CONDITIONS: Infertility
Keywords: IVF; embryos; research; donation; surplus; stem cells
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Biospecimen Retention: Samples With DNA — Blood serum samples of donor couple. Reproductive samples of donor couple
  Note: number of subjects indicates 40 donor couples (40 x 2 = 80 subjects)
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Human embryonic stem cells (hESCs) are isolated from the early human embryo and have the capability to proliferate indefinitely in culture and to develop into nearly every cell of the human body. Therefore, hESCs may serve as a renewable unlimited source of cells for transplantation therapy. Because of the use of animal products in their derivation, and due to the lack of appropriate quality and process controls in the manufacturing of existing cell lines worldwide, existing hESC lines are not suitable for utilization in transplantation therapy.

Our objective is to derive several new hESC lines that will be suitable for clinical trials. The investigators plan on deriving the new hESC lines utilizing only FDA-approved raw materials in a non-animal culture system. They will be produced entirely under GMP conditions, using appropriately documented procedures and analytical methods, completely safety tested, and screened for infectious and adventitious agents.

DETAILED DESCRIPTION:
Embryonic stem (ES) cell lines are derived from the pluripotent cells of the early embryo. The key properties of ES cells are their ability to proliferate indefinitely in vitro without differentiation, and their capability to give rise to all cells of the body. The recent derivation of ES cell lines from human embryos (Thomson et al., 1998, Reubinoff et al., 2000) attracts significant attention due to the remarkable potential of these cells for basic scientific research, drug development, and regenerative medicine.

Since human embryonic stem cells (hESCs) are capable of unlimited self-renewal and can give rise to any specialized cell via differentiation, they can potentially be used as an unlimited donor source of cells for transplantation in a variety of disorders that result from the loss of cells or cellular dysfunction. Among these conditions is Parkinson's disease, multiple sclerosis, traumatic spinal cord injury, diabetes, heart failure, liver failure, etc.

It has been proposed that the essential characteristics of primate ES cells should include (i) derivation from the preimplantation or periimplantation embryo, (ii) prolonged undifferentiated proliferation, and (iii) stable developmental potential to form derivatives of all three embryonic germ layers even after prolonged culture (Thomson, 1996). The investigators have derived stem cell lines from early human embryos that meet these criteria (Reubinoff et al., 2000). Our group was second in the world to derive hESC lines, and the first to show their potential to undergo somatic differentiation in vitro (Reubinoff et al., 2000).

To exploit the remarkable potential of hESCs, improvement of currently used methods for culturing and manipulating the cells as well as controlling their differentiation are required. In this context, the investigators have developed novel approaches to cryopreserve (Reubinoff et al., 2001), to genetically modify (Gropp et al., 2003; Ben-Dor et al., 2006) and to control the differentiation of hESCs cells (Reubinoff et al., 2001, Itsykson et al., 2005).

Human ES cell lines are derived from embryos produced by in vitro fertilization (IVF) for clinical purposes. Surplus frozen embryos that are no longer required for infertility treatment are recruited for this purpose after donor informed consent and institutional/national review board approvals are obtained. The embryos are thawed and cultured to the blastocyst stage (5-6 days), the inner cell mass (ICM) comprised of pluripotent cells is isolated, and the stem cells are most commonly cultured on mouse embryonic fibroblast feeder cell layer. The feeder layer is required to prevent differentiation and to promote the proliferation of the stem cells.

Most hESC lines reported worldwide to date and all the cell lines currently listed in the NIH registry were derived on mouse fibroblast feeder layers. The current lines would not be suitable for clinical use, as the screening of donors and reagents was not FDA compliant, and the presence of the mouse feeders renders these lines xenotransplantation products. The regulatory compliance issues these lines raise make it difficult to obtain FDA approval for human transplantation use.

To eliminate the use of mouse feeders, undifferentiated hESCs can be successfully propagated on laminin or Matrigel-coated plastic surfaces in the presence of mouse embryonic fibroblast-conditioned medium (Xu et al 2001). While this system avoids direct contact between mouse feeders and hESCs, the risk of cross-transfer of animal pathogens from the animal-conditioned medium to the hESCs is not avoided. During the early days of developing our cell lines, the investigators successfully cultivated the hESCs on human feeders. Subsequently, Richards and his colleges demonstrated that human fetal and adult feeders support prolonged undifferentiated propagation of existing hESC lines and are superior to cell-free matrices supplemented with human or mouse feeder-conditioned medium. They also reported the derivation of a new hESC line using human embryonic fibroblasts and animal-free culture conditions (Richards et al., 2002). The potential use of human placenta and foreskin-derived feeders to develop and support undifferentiated propagation of hESCs was also demonstrated (Genbacev et al., 2005; Amit et al., 2003).

Maintenance of cultures of undifferentiated hESCs in the absence of feeders was recently reported. It was shown that the combination of LIF, basic fibroblast growth factor, and transforming growth factor Beta1 can support undifferentiated proliferation of hESCs on fibronectin (Amit et al., 2004). The activation of the Wnt signaling system was also suggested to promote the maintenance of pluripotent hESCs in the absence of feeders (Sato et al., 2004). Furthermore, it has been suggested that substituting the medium with high concentrations of FGF2 and noggin is sufficient to support the propagation of hESCs without feeders (Xu et al., 2005). In addition, feeder-free undifferentiated propagation of hESCs colonies was reported with a chemically-defined medium without serum replacer, supplemented with activin or nodal plus FGF2 (Vallier er al., 2005). Lastly derivation and propagation of hESCs in an animal free, chemically-defined, feeder-free culture system in the presence of high concentrations of FGF2 was reported (Ludwig et al., 2006). So far, the development of hESC under conditions that will allow there future use for transplantation therapy was not reported.

In the second half of the project, the investigators propose to continue our efforts to develop new clinical-grade hESC lines derived totally from FDA-approved raw materials in a non-animal culture system.

The mouse feeders will be replaced with primary cell lines of human fibroblasts. In the first part of the project, the investigators have completed the development of master cell banks (MCBs) of clinical-grade human fibroblast feeders. These feeders were produced entirely under GMP conditions within the Hadassah Vector Production Facility, using animal-free, FDA-approved raw materials (for details see Results section). To the best of our knowledge, the development of GMP clinical-grade human feeders was not reported by other groups.

In parallel, the investigators have modified the methods for the derivation and culture of hESCs. The investigators have developed novel animal-free methods for the isolation of the pluripotent stem cells from human IVF embryos and successfully used these methods in the derivation of new hESC lines. The replacement of animal products and FDA non-approved materials with humanized or recombinant clinical-grade materials in the hESC culture system is near completion. Validation of the efficacy of the modified culture system is ongoing. Preliminary results suggest that the modified culture system can efficiently support undifferentiated cultivation of hESCs.

The newly-derived clinical-grade hESC lines will be derived using embryos from couples entirely screened according to organ donation and blood donation guidelines and regulations (per the FDA proposed rule for donor suitability). In the first year, the investigators have completed the recruitment of 14 embryos from three couples. Donor medical histories were reviewed, and screening blood and swab test results were obtained and documented. Samples of donor couple blood were archived for retrospective testing in a locked storage facility. Recruitment of additional embryos is ongoing.

Upon completion of the characterization and safety testing of the new human feeders, expanding them into working lots, and validation of the efficacy of the clinical grade-culture system for hESCs, the investigators will develop the new hESC lines in the Hadassah University Hospital Vector Production Facility, whereby stringent quality control and environmental testing will be maintained. All work will be accomplished utilizing only raw materials approved by our Quality Assurance Program, provided by vendors who underwent a strict vendor approval/review process. The production work will be performed using techniques adhering to good manufacturing practices (GMPs) and good tissue practices (GTPs).

Early passage hESCs and feeders (Master Cell Bank) will be submitted for phenotypic and latent agent testing, endotoxin analysis, and testing for viral and adventitious agent contamination. The Working Cell Bank of both feeders and hESCs will be also tested for phenotypic characterization, reproducibility, sterility, and mycoplasma, detection of latent agents, and endotoxins. The final product will be retested as per the Master Cell Bank, above.

By the conclusion of our manufacturing and testing process, Hadassah's Stem Cell Program will provide a generic commercial product. The procedures and methods that the investigators have developed will be instrumental tools to other stem cell researchers, thus paving the way for the future of stem cell research in Israel and worldwide. The commercial potential of the product will allow production of specific cells for clinical use; they will have a widespread commercial value and will be of enormous market worth.

ELIGIBILITY:
Inclusion Criteria:

* Couple has embryos derived through IVF that they wish to donate to research.
* Couple has finished building their family.
* Couple has them stored in liquid nitrogen for > or = to 5 years.
* Couple will submit to an interview, blood tests, and physical exam by a physician.
* Couple will give informed consent and will consent to have their medical history examined by the research group.

Exclusion Criteria:

* Couple has not finished building their family.
* Couple has embryos but they have not been stored for > or = to 5 years.
* Couple will not submit to an interview, blood tests, or physical exam by a physician.
* Couple refuse to give informed consent, or will not consent to have their medical history examined by the research group.
* Couple has spent an extended period of time in exclusion countries (HIV or vCJD risk).
* Couple tests positive for exclusion viruses (as listed in the Informed Consent).

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Embryo donors who have derived embryos via IVF and have surplus embryos that they will not use for family-building.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2002-07-07 (Actual); Primary Completion 2030-12 (Estimated); Study Completion 2030-12 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin E. Reubinoff, M.D. PhD., Principal Investigator — Hadassah Medical Organization
Locations (1):
- Hadassah Medical Organization, Jerusalem, Israel

REFERENCES:
- [Background] Reubinoff BE, Pera MF, Fong CY, Trounson A, Bongso A. Embryonic stem cell lines from human blastocysts: somatic differentiation in vitro. Nat Biotechnol. 2000 Apr;18(4):399-404. doi: 10.1038/74447. PMID 10748519
- See also: Link to Hadassah's Human Embryonic Stem Cell Research Center — https://www.hhesc.co.il